CLINICAL TRIAL: NCT04951141
Title: Beijing Immunochina Medical Science & Technology Co., Ltd.
Brief Title: Clinical Study of Intratumoral Injection of CAR-T Cells in the Treatment of Advanced Liver Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-003-D
Record Dates: First submitted 2021-06-24; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Hepatocellular Carcinoma , Cholangiocarcinoma
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-GPC3 CAR-T (Experimental)
  Interventions: Biological: anti-GPC3 CAR-T cells

INTERVENTIONS:
Biological: anti-GPC3 CAR-T cells — A single arm, open-label pilot study is designed to determine the safety and efficacy of anti-GPC3 CAR-T cells in patients with GPC3-positive advanced liver cancer.

SUMMARY:
Objective to study the safety and preliminary efficacy of intratumoral injection of CAR-T cells in the treatment of advanced liver tumors.

ELIGIBILITY:
Inclusion Criteria:

* GPC3 expression was positive by histological examination;
* 18-69 years old;
* The patients with advanced liver tumor who can not be operated and the effect of chemotherapy is poor;
* The patients who received traditional palliative therapy had an expected survival period of more than 4 months;
* Organ status allows clinical application.a. Creatinine < 1.5mg/dl; b. Cardiac ejection index > 55%; c. Heme > 9g / dl, bilirubin < 2.0mg/dl;
* No bleeding and coagulation disorders were found;
* There was no allergy to contrast medium;
* Contraception: contraceptive measures were taken during clinical application and within 3 months after the last cells transfusion;
* There is no other contraindication for lymphocyte collection;
* Sign informed consent.

Exclusion Criteria:

* Pregnant or lactating women;
* Patients need systemic steroids therapy;
* At present, the treatment conditions are as follows : a. Within 30 days before the collection of peripheral blood mononuclear cells,patiens were in other anti-tumor clinical observation period; b. Patients have not recovered from the acute side effects of previous treatment;
* Patients received radiotherapy within 4 weeks after enrollment;
* Patients received other cell modification therapy in the early stage;
* In the screening stage, patients with lymphocyte transfection rate less than 5%, or T cell culture can not expand (< 5 times) patients;
* Uncontrolled symptoms or other diseases include, but are not limited to, infection, congestive heart failure, unstable angina pectoris, arrhythmia, psychosis, or limiting the social environment that meets the requirements, or the researchers believe that they may bring unpredictable risks;
* Patients with severe acute allergic reactions;
* Patients who participated in other clinical trials;
* Researchers believe that patients are not suitable to participate.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
Adverse events attributed to the administration of the anti-GPC3 CAR-T cells | 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
Overall survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yin ying Lu, M.D., Principal Investigator — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of Chinese PLA General Hospital, Beijing, China